CLINICAL TRIAL: NCT04456374
Title: Evaluation of Soccer-specific Performance and Body Composition in Youth Soccer Players of Different Age Groups
Brief Title: Performance Testing in Young Soccer Players
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Other Study IDs: YOUTH SOCCER STUDY-UTH-2020
Record Dates: First submitted 2020-06-24; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Physical Performance
Keywords: soccer; performance; youth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Under-12 (U12) players
  Interventions: Other: Performance testing
- Under-14 (U14) players
  Interventions: Other: Performance testing
- Under-16 (U16) players
  Interventions: Other: Performance testing
- Under-18 (U18) players
  Interventions: Other: Performance testing

INTERVENTIONS:
Other: Performance testing — Soccer-specific performance will be evaluated by measuring flexibility, jumping ability, maximum speed, repeated spring ability, agility and endurance.

SUMMARY:
The aim of this study is to investigate physiological characteristics, body composition and performance indicators among youth soccer players of four age categories (U-12, U-14, U-16, and U-18). Participants will undergo assessment of their body weight, body height and percent of body fat as well as performance testing including flexibility, strength, vertical jump, speed, repeated sprint ability, agility, dribbling and endurance.

DETAILED DESCRIPTION:
This study aims at investigating anthropometric, body composition and performance indicators among male youth soccer players. The study will be conducted prior to the preparation period. Initially, participants and their parents (for those under 18 years) will be informed about the benefits, risks and discomforts associated with the study and will provide a written consent. Participants will be instructed to refrain from strenuous exercise for at least 48 hours prior to testing and they will be also asked to consume their normal diet. Prior to testing all participants will be familiarized with testing procedures and specific test. Body weight will be measured on a seca beam balance. Participants' height will be measured by using a fixed stadiometer and the percent body fat will be calculated with bioelectrical impedance analysis. Flexibility will be assessed by using the sit and reach test and the lower body explosive strength will be determined through vertical jump testing (squat jump and counter movement jump without arm swing). Knee flexor and extensor strength will be assessed on an isokinetic dynamometer. Sprint performance will be assessed from a standing start over by infrared photocells with participants running 10m and 30m as fast as they can. The repeated sprint ability will be tested by using linear sprint test including 5 maximum sprints of 30 meters with a 25-second recovery period in-between. Maximal oxygen consumption (VO2max) will be determined by open-circuit spirometry via breath-by-breath analysis during a graded exercise test to exhaustion on a treadmill. Furthermore, participants will be evaluated in agility by using the short dribbling test and the ability to recover after repeated intense exercise through the YO-YO Intermittent Recovery test 1 (only for u-16 and U-18 groups).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 11 and 12 years
* Active soccer players participating in regular soccer practice and competition
* Training age ≥ 3 years
* Free of chronic diseases
* Free of musculoskeletal injury

Exclusion Criteria:

* Musculoskeletal injury
* Chronic disease
* Training age ≤ 2 years

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Youth soccer players (aged 11-18 years) participating in regular soccer practice and competition with a training age of ≥ 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-08-05 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
Flexibility | At baseline
  Flexibility will be assessed by using the sit-and-reach test
Jumping ability | At baseline
  Jumping ability will be assessed by measuring the vertical jumping performance using two different techniques: i) countermovement and ii) squat jump.
Maximum speed | At baseline
  Maximum speed will be assessed over 10 m and 30 m by using light cells
Repeated sprint ability | At baseline
  Repeated sprint ability will be assessed by performing five 30-m sprints with 25 seconds recovery period in-between, and using light cells.
Agility | At baseline
  The ability to change direction while dribbling the ball (termed agility) will be assessed by using the short dribbling test (performed according to standard procedures).
Endurance | At baseline
  Endurance will be assessed by using the Yo-Yo Intermittent Recovery test level 1
Maximal oxygen consumption (VO2max) | At baseline
  Maximal oxygen consumption will be measured by open-circuit spirometry via breath-by-breath analysis during a graded exercise test to exhaustion on a treadmill, using automated pulmonary gas exchange system.
Knee flexor and extensor strength | At baseline
  Concentric and eccentric peak torque of knee flexors and extensors in both limbs (dominant and non-dominant) will be assessed on an isokinetic dynamometer

SECONDARY OUTCOMES:
Body height | At baseline
  Body height will be measured on a beam balance with stadiometer.
Body weight | At baseline
  Body weight will be measured on a beam balance with stadiometer.
Body composition | At baseline
  Body fat and fat-free mass will be estimated by using bioelectrical impedance.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Poulios, PhD, Principal Investigator — University of Thessaly
Locations (1):
- University of Thessaly, School of Physical Education and Sports Science, Trikala, Greece

IPD SHARING:
Plan to Share IPD: Undecided